CLINICAL TRIAL: NCT02036892
Title: Electronically Connected Health Coaching in Improving Type 2 Diabetes Self Management - Phase III Trial
Brief Title: Electronically Connected Health Coaching in Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: York University (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Paul Ritvo, Associate Professor, School of Kinesiology and Health Science, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-001
Record Dates: First submitted 2014-01-06; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling with smartphones (Experimental): Lifestyle counseling assisted by smartphones
  Interventions: Behavioral: Lifestyle counseling with smartphone
- Lifestyle counseling (Active Comparator): Lifestyle counseling
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling with smartphone — Lifestyle counseling with health promoting smartphone software
  Arms: Lifestyle counseling with smartphones
Behavioral: Lifestyle counseling — Lifestyle counseling
  Arms: Lifestyle counseling

SUMMARY:
Patients with Type 2 Diabetes randomly allocated to the intervention arm (health coaching + smartphone-based health promotion software) will have significantly better Hemoglobin A1c levels at 6 months post-intervention than patients with Type 2 Diabetes allocated to the control arm (health coaching alone).

DETAILED DESCRIPTION:
Inclusion criteria: all participating patients have been diagnosed with Type 2 Diabetes, are between 25 and 70 years of age, have a regular primary care physician, and have HbA1c levels > or = to 7.3.

Exclusion criteria: Axis I and II psychiatric disorders.

Primary outcome: HBA1c at 6 months follow up.

Secondary outcome: Centre for Epidemiological Studies Depression Scale

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes
* Fluency in English and/or Spanish

Exclusion Criteria:

* > 75 years of age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 months follow up from baseline
  Finger prick A1c test or lab test

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale | 6 months follow up from baseline assessment
  Self report measure of psychological distress

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ritvo, PhD, Principal Investigator — York University
Locations (1):
- Black Creek Community Health Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wayne N, Perez DF, Kaplan DM, Ritvo P. Health Coaching Reduces HbA1c in Type 2 Diabetic Patients From a Lower-Socioeconomic Status Community: A Randomized Controlled Trial. J Med Internet Res. 2015 Oct 5;17(10):e224. doi: 10.2196/jmir.4871. PMID 26441467
- [Derived] Pludwinski S, Ahmad F, Wayne N, Ritvo P. Participant experiences in a smartphone-based health coaching intervention for type 2 diabetes: A qualitative inquiry. J Telemed Telecare. 2016 Apr;22(3):172-8. doi: 10.1177/1357633X15595178. Epub 2015 Jul 21. PMID 26199275